CLINICAL TRIAL: NCT02418221
Title: A Doubleblind, Placebo-controlled, Cross-over Provocation Study Using Biogenic Amines to Show the Efficacy of Oral Diamine Oxidase (DAOSiN®) Supplementation in Case of DAO Enzyme Deficiency
Brief Title: A Provocation Study Using Biogenic Amines to Show the Efficacy of Oral Diamine Oxidase Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IPSC AG (Industry)
Collaborators: Medical University of Graz (Other); Sciotec Diagnostic Technologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Provokamin01
Record Dates: First submitted 2014-09-01; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Histamine Intolerance
Keywords: histamine, biogenic amines, diamine oxidase
MeSH Terms: interventions — Pulse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DAOSiN®/ Placebo & ProvokAmin® Ingestion (Experimental): A sample of blood is drawn from Patient, blood pressure & pulse are recorded. Patient will ingest 2 capsules of either DAOSiN® or Placebo, followed by 2 tablets of ProvokAmin 20 minutes later. After an additional 40 minutes blood pressure and pulse are recorded and another sample of blood is drawn. Patient is handed a questionaire for self-evaluation to record any symptoms for the following After between 7 and 15 days the whole cycle is repeated switching between active treatment and Placebo.
  Interventions: Dietary Supplement: DAOSiN®/ Placebo & ProvokAmin® Ingestion; Procedure: Drawing blood, measuring BP & pulse

INTERVENTIONS:
Dietary Supplement: DAOSiN®/ Placebo & ProvokAmin® Ingestion — Proband is randomly assigned Daosin® or the Placebo before provocation with ProvokAmin®
Procedure: Drawing blood, measuring BP & pulse — Taking of a blood sample and recording of blood pressure & pulse

SUMMARY:
This study aims to define a provocation test for histamine intolerance (aka. biogenic amine intolerance syndrome) and test the capability of an oral enzyme supplementation to ameliorate this condition.

DETAILED DESCRIPTION:
The clinical picture of the so-called histamine intolerance has been described by various authors since the 1990ies. However, the existence of this multifactorial condition is also being contested due to the lack of both a positive definition and unambiguous diagnostics. Various provocation studies using pure histamine or histamine-containing foods support the existence of the disease pattern, however many questions still remain open.

A lack of diamine oxidase (DAO) is considered the etiological cause of the condition. DAO is an enzyme known to degrade a wide array of biogenic amines. The aim of this study is to provoke a response in patients by oral administration of a defined mixture of biogenic amines. By administration of DAO before provocation an attenuation of the symptoms is to be expected.

ELIGIBILITY:
Inclusion Criteria:

* Persons suspected of suffering from BAIS (BAIS Score ≥ 50) according the the questionaire used for histamine intolerance so far

Exclusion Criteria:

* pregnancy
* coronary heart disease
* labile hypertension
* bronchial asthma
* periodical therapy using H1-blockers
* chirurgical intervention with the GI tract within the previous 3 months
* participation in a clinical trial within the previous 4 weeks

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Reduction of biogenic amine symptoms (determined via symptom score) | 24 hrs after start of provocation
  The primary parameter is the reduction of clinical symptoms caused by the ingestion of biogenic amines by the preventive oral administration of DAOSiN®. A symptom score quantifying the subjective single symptoms is used as measuring parameter.

SECONDARY OUTCOMES:
Serological parameters | Up to 90 min after provocation
  These parameters are ascertained: DAO activity and concentration of histamine in serum; blood pressure & pulse measurement before and 30/60/90 min post provocation

CONTACTS AND LOCATIONS:
Overall Officials: Albert Missbichler, PhD, Study Chair — Sciotec Diagnostic Technologies GmbH
Locations (1):
- Department of Environmental Dermatology and Venereology, Medical University of Graz, Graz, Austria